CLINICAL TRIAL: NCT04663763
Title: The Combination of Neoadjuvant Short-course Radiotherapy and Immunotherapy in Locally Advanced Rectal Cancer：A Open-label Single-arm Phase II Trial.
Brief Title: Neoadjuvant Short-course Radiotherapy Followed by the Combination of Immunotherapy and Chemotherapy in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-336
Record Dates: First submitted 2020-11-28; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant short-course radiotherapy; Immunotherapy; Locally advanced rectal cancer; Pathological complete response
MeSH Terms: interventions — spartalizumab; sintilimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant short-course radiotherapy+immunotherapy+chemotherapy (Experimental): A total of 40 patients receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody, finally receive the TME surgery and another 4 cycles of CAPOX chemotherapy.
  Interventions:
  Shor-course radiotherapy: 25Gy/5Fx;
  Induction immunotherapy: Sintilimab 200mg ivgtt d1 q3w x 4 cycles;
  Concurrent Chemotherapy: Oxaliplatin: 130mg/m2 d1 q3w + Capecitabine: 1000mg/m2 d1-14 q3w x 4 cycles;
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: PD-1 antibody — Sintilimab is a humanized IgG4 monoclonal antibody against the programmed death-1 (PD-1) receptor. Usage: 200mg ivgtt d1 q3w.
  Other Names: Sintilimab
Drug: Capecitabine — Usage: 1000mg/m2 d1-14 q3w
Drug: Oxaliplatin — Usage: 130mg/m2 d1 q3w

SUMMARY:
This is a single arm, open-label, prospective phase II clinical trial to evaluate the combination of neoadjuvant short-course radiotherapy and immunotherapy (PD-1 antibody) for patients with locally advanced rectal cancer (LARC). A total of 40 patients will be enrolled in this trial to receive 5*5Gy short-course radiotherapy, followed by 4 cycles of CAPOX chemotherapy and PD-1 antibody. Then they will receive the TME surgery and another 4 cycles of CAPOX chemotherapy. There are two cohorts according to the microsatellite instability status: (1) the micro-satellite stable (MSS) cohort（n=32), (2) the MSI-high cohort (n=8). The primary end point is the rate of pathological complete response (pCR). The long-term prognosis and adverse effects will also be evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathological confirmed rectal adenocarcinoma and the distance from anal verge less than 12 cm;

  2. Clinical stage T3-4 and/or N+ (AJCC 8th);

  3. No distant metastases;

  4. Age 18-70 years old, female and male;

  5. ECOG 0-1;

  6. No previous chemotherapy, radiotherapy, immunotherapy or other anti-tumor treatment;

  7. Adequate organ function defined at baseline as:
  1. ANC ≥1.5×109 /L，PLt ≥75×109 /L，Hb ≥90 g/L;
  2. TBIL ≤1.5×ULN, ALT ≤2.5ULN, AST ≤2.5ULN, BUN and Cr ≤1×ULN or Ccr ≥50ml/min (Cockcroft-Gault formula);
  3. INR ≤1.5×ULN or PT ≤1.5×ULN (If the patient is receiving anticoagulant therapy, PT should be within the intended use range of the anticoagulant drug);

  8. With good compliance and no serious comorbidity;

  9. Women of childbearing age must have taken reliable contraceptive measures or have a pregnancy test (serum or urine) within 7 days prior to enrollment and the results are negative;

  10. Subject volunteers to join the study, sign the informed consent.

Exclusion Criteria:

* 1. History of other uncured malignancies within 5 years. Cured tumor with good prognosis, such as skin basal cell carcinoma, cervical cancer and superficial bladder cancer, will be excluded;

  2. Have received surgery within 4 weeks before the enrollment;

  3. History of obstruction within 6 months before the enrollment;

  4. History of active autoimmune disease, interstitial lung disease, epilepsy and dysphrenia;

  5. With uncontrolled cardiovascular disease: active coronary heart disease; grade III-IV cardiac insufficiency according to the NYHA criteria; and myocardial infarction within 1 year;

  6. With active infection or fever of >38.5 ℃ with unknown cause (tumor-induced fever judged could be enrolled);

  7. DPD deficiency;

  8. Allergic to any component of chemotherapy or immunotherapy;

  9. With congenital or acquired immunodeficiency (such as those with HIV infection), active hepatitis B or hepatitis C;

  10. Usage of corticosteroids (prednison dose of > 10 mg/day) or other immunosuppressors for systemic treatment within the first 14 days of research;

  11. Receive attenuated live vaccine within 4 weeks before the research;

  12. Pregnant women or breast-feeding women;

  13. With other factors that would force to terminate the clinical trial ahead of time, such as the development of other severe comorbidity that required combined treatment, and family or social factors affecting the safety of patients or experimental data collection, as judged by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | The TME surgery will be recommended at 1 week after the neoadjuvant therapy. The pCR rate is evaluated after surgery. Assessed up to 6 months
  Pathologic complete response rate

SECONDARY OUTCOMES:
3-year DFS | Assessed up to 3 years
  3-year disease free survival rate
3-year local recurrence rate | Assessed up to 3 years
  3-year local recurrence rate
3-year OS | Assessed up to 3 years
  3-year overall survival rate
Grade 3-4 adverse effects rate | Assessed up to 3 years
  Radiotherapy, immunotherapy and chemotherapy related grade 3-4 adverse events rate
Surgical complications | Assessed up to 3 years from the TME surgery
  Type and Rate of surgical complications
Quality of Life Scale | Assessed up to 5 years
  The Quality of Life Scale (QoLS, range 0-60) will be used to evaluate the quality of life. Higher scores mean the better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Zhu, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No